CLINICAL TRIAL: NCT00795119
Title: A Clinical Assessment of the Reliability of Near Infrared Spectroscopy for the Detection of Intracranial Hemorrhage in Young Children
Brief Title: A Trial to Determine the Efficacy of Near Infrared Spectroscopy to Detect Intracranial Hemorrhage in Children
Acronym: NIRS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IWK Health Centre (Other)
Responsible Party: Dr Steven Bellemare, IWK Health Centre, Dalhousie University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IWK3748
Record Dates: First submitted 2008-11-19; First posted 2008-11-21 (Estimated); Last update posted 2009-04-03 (Estimated); Status verified 2008-11

CONDITIONS: Intracranial Hemorrhage
Keywords: Near Infrared Spectroscopy; Diagnosis; Children
MeSH Terms: conditions — Intracranial Hemorrhages; Disease | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NIRS (Experimental): Children who undergo NIRS
  Interventions: Device: Near Infrared Spectroscopy (NIRS)

INTERVENTIONS:
Device: Near Infrared Spectroscopy (NIRS) — NIRS of the head is undertaken at the time of CT or MRI examination

SUMMARY:
To diagnose bleeding inside the head, children need to have a CT Scan or MRI of their heads. Not all doctors order these though, especially when there is no history of injury or when children don't look too sick. Unfortunately, this means that some children's bleeding doesn't get diagnosed as early as it could. This study wants to find a way to detect bleeding inside the head without using a CT scan or MRI.

ELIGIBILITY:
Inclusion Criteria:

* All children under 3 years of age who undergo a CT of the head or MRI of the head.

Exclusion Criteria:

* Lack of parental consent
* Neurosurgical intervention between CT/MRI and NIRS scanning.
* Scalp hematoma

Max Age: 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2007-09; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Sensitivity of NIRS | Study conclusion

SECONDARY OUTCOMES:
specificity of NIRS, positive/negative predictive value | Study conclusion

CONTACTS AND LOCATIONS:
Overall Officials: Steven Bellemare, MD, Principal Investigator — IWK Health Centre
Locations (1):
- IWK Health Centre, Halifax, Nova Scotia, Canada